CLINICAL TRIAL: NCT05245175
Title: Assessment of Impact of Different Carrier Solutions for House Dust Mite Allergen (HDM) Challenge on Allergic Reactions in Patients with HDM Allergic Rhinitis
Brief Title: Impact of Carrier Solutions for House Dust Mite Allergen on Allergic Reactions
Acronym: SIMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jens Hohlfeld, MD, Division Director of Airway Research, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 22-05 SIMBA
Record Dates: First submitted 2022-01-26; First posted 2022-02-17 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2022-07

CONDITIONS: Allergic Rhinitis
Keywords: Allergen Challenge Chamber; House dust mite; Sodium chloride
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Environment, Controlled; Antigens, Dermatophagoides

STUDY DESIGN:
Intervention Model Description: 18 patients will be exposed 5 times in the Allergen Challenge Chamber. The 5 exposures are divided into 2 blocks. The first block consists of 3 challenges with sodium chloride particles, lactose particles, and clean air to address the primary and secondary objectives. The second block consists of 2 further challenges with D. pteronyssinus coupled with either sodium chloride particles or lactose particles to address exploratory objectives.
Who Masked: Participant
Masking Description: Patients are blinded to the sequence of exposures. Within the 2 blocks, the order of challenge atmospheres will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Sodium chloride particles (Experimental): Patients are exposed to sodium chloride particles alone for 4 hours in the Fraunhofer Allergen Challenge Chamber.
  Interventions: Other: Sodium chloride particles
- Lactose particles (Experimental): Patients are exposed to lactose particles alone for 4 hours in the Fraunhofer Allergen Challenge Chamber.
  Interventions: Other: Lactose particles
- Clean air (Placebo Comparator): Patients are exposed to clean air for 4 hours in the Fraunhofer Allergen Challenge Chamber.
  Interventions: Other: Clean air
- Sodium chloride particles with house dust mite (Experimental): Patients are exposed to sodium chloride particles coupled with D. pteronyssinus for 4 hours in the Fraunhofer Allergen Challenge Chamber.
  Interventions: Other: Sodium chloride particles with house dust mite
- Lactose particles with house dust mite (Experimental): Patients are exposed to lactose particles coupled with D. pteronyssinus for 4 hours in the Fraunhofer Allergen Challenge Chamber.
  Interventions: Other: Lactose particles with house dust mite

INTERVENTIONS:
Other: Sodium chloride particles — Patients are exposed to sodium chloride particles alone for 4 hours in the Fraunhofer Allergen Challenge Chamber.
  Arms: Sodium chloride particles
Other: Lactose particles — Patients are exposed to lactose particles alone for 4 hours in the Fraunhofer Allergen Challenge Chamber.
  Arms: Lactose particles
Other: Clean air — Patients are exposed to clean air for 4 hours in the Fraunhofer Allergen Challenge Chamber.
  Arms: Clean air
Other: Sodium chloride particles with house dust mite — Patients are exposed to sodium chloride particles coupled with D. pteronyssinus for 4 hours in the Fraunhofer Allergen Challenge Chamber.
  Arms: Sodium chloride particles with house dust mite
Other: Lactose particles with house dust mite — Patients are exposed to lactose particles coupled with D. pteronyssinus for 4 hours in the Fraunhofer Allergen Challenge Chamber.
  Arms: Lactose particles with house dust mite

SUMMARY:
Single-blind, within-block randomized, clean-air-controlled study to assess the effect of lactose and sodium chloride particles in patients with allergic rhinitis on nasal symptoms when challenged in the Fraunhofer Allergen Challenge Chamber

DETAILED DESCRIPTION:
Allergen Challenge Chambers (ACC) are used worldwide since many years to test anti-allergic treatment in early clinical development. ACCs provide the advantage of controlled atmospheres with stable allergen load and highly reproducible symptoms during challenges.

The Fraunhofer ACC has been used since more than 20 years to test a range of different anti-allergic treatments, mostly using pollen challenges.

For house dust mite (HDM) challenges, a carrier solution containing lactose or sodium chloride is reconstituted with commercially available HDM allergen. The solution is spray-dried to create allergen loaded lactose or sodium chloride particles of a determined size. Those particles are distributed in the ACC.

Whether lactose or sodium chloride particles alone could induce nasal irritation during allergen challenges, has not been examined. Should allergen-free carrier solutions contribute to nasal symptoms, study results might be confounded. Even more so, if one carrier solution caused more nasal irritation than the other.

To determine if allergen-free carrier solutions alone irritate the nasal mucosa, we expose subjects with allergic rhinitis and house dust mite allergy to three different atmospheres: (1) lactose particles alone, (2) sodium chloride particles alone, and (3) clean air. Also, we aim to document nasal symptoms during challenges with HDM-containing carrier solutions to decide on the best carrier option for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent.
2. Male and female subjects, aged 18-65 years. Women will be considered for inclusion if they are:

   * Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing.
   * Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).
   * Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first allergen challenge until at least 72 hours after the last allergen challenge -, implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).
3. Body mass index between 18 and 32 kg/m2
4. History of HDM-induced allergic rhinitis with or without conjunctivitis of 1 year or longer in duration at screening.
5. Positive skin prick test responses (positive wheal diameter reaction of ≥ 3 mm larger than the negative control and wheal diameter < 2 mm to the sodium chloride/diluent negative control) to D. pteronyssinus at screening or within the past 12 months (if performed and documented at the clinical unit).
6. Serum specific IgE level (≥ 0.7 kU/L) to D. pteronyssinus at screening or within the past 12 months (if performed and documented at the clinical unit).
7. FEV1 of 80% of predicted value or greater at screening. If subject fails to achieve this value, the assessment may be repeated 2 additional times.
8. Total Nasal Symptom Score (TNSS) of ≤ 3 prior to entering the chamber at visit 2.
9. Smokers or non-smokers.

Exclusion Criteria:

1. Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urine analysis, vital signs, lung function or ECG at screening visit , which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study, or the subject's ability to participate in the study.
2. Diastolic blood pressure above 95 mmHg.
3. Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
4. History of an acute infection at screening that has not resolved four weeks prior to visit 2.
5. Nasal condition that could confound the efficacy or safety assessments (e.g., nasal polyps).
6. Concomitant allergies to seasonal aeroallergens which are anticipated to be or become active (i.e., grass, trees, weeds, rye; defined as IgE ≥ 3.5 kU/L [IgE samples drawn within 12 months prior to screening can be used to assess criteria as long as they are performed and documented at the clinical unit]; OR symptomatic to aeroallergens within the past 2 years or within the past 2 allergy seasons; OR both) through the completion of the study.
7. Concomitant allergy to an animal dander who has exposure on a regular basis to the respective animal dander.
8. History of allergic reactions such as anaphylactic shock, exanthema generalized, angioedema or hypotension caused by HDM and/or any medical products (including vaccine) in the past.
9. Known or suspected clinically relevant intolerance to lactose .
10. Asthma other than mild asthma which is treated with short acting beta-2-agonists only and which is controlled according to the current GINA guidelines.
11. Participation in another clinical trial 30 days prior to enrollment.
12. Donation of more than 400 ml of blood the preceding 2 months before screening.
13. History of regular drug or alcohol abuse in the past 3 months.
14. Risk of non-compliance with study procedures.
15. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
16. Specific Immunotherapy (SIT) within five years prior to the study.
17. Treatment with medication that might interfere with rescue medication for anaphylactic reactions (e.g. beta blocker).
18. Systemic immunosuppression treatment (e.g. oral steroids, biologics, e.g. dupilumab, JAK-Inhibitors, cyclosporine, azathioprine, Mycophenolat Mofetil (MMF) within 3 months before visit 2
19. Treatment with anti-allergic medication or topical steroids (within 2 weeks before visit 2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Change of mean total nasal symptom score (TNSS) during challenge over 4 hours with either lactose or sodium chloride particles compared to challenges with clean air. | Day 1, Day 2, Day 3
  TNSS = Total Nasal Symptom Score (min = 0 = no symptoms; max = 12 = max symptoms)

SECONDARY OUTCOMES:
Change of mean VAS of symptoms during challenge over 4 hours with either lactose or sodium chloride particles compared to challenges with clean air | Day 1, Day 2, Day 3
  VAS = Visual Analogue Scale (min = 0 = no symptoms; max = 10 = max symptoms)
Difference in nasal secretion weight during challenge over 4 hours with either lactose or sodium chloride particles compared to challenges with clean air | Day 1, Day 2, Day 3
  Pre-weighed handkerchief sachets used by subjects during challenge are weighed after use to determine nasal secretion amount

OTHER OUTCOMES:
Change of mean total nasal symptom score (TNSS) during challenge over 4 hours with either HDM allergen with lactose particles compared to challenges with HDM allergen with sodium chloride particles. | Day 4, Day 11
  TNSS = Total Nasal Symptom Score
Change of nasal secretion weight during challenge over 4 hours with either HDM allergen with lactose particles compared to challenges with HDM allergen with sodium chloride particles | Day 4, Day 11
  Pre-weighed handkerchief sachets used by subjects during challenge are weighed after use to determine nasal secretion amount

CONTACTS AND LOCATIONS:
Overall Officials: Jens M Hohlfeld, Prof. Dr., Principal Investigator — Fraunhofer Institute for Toxicology and Experimental Medicine ITEM
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lueer K, Biller H, Casper A, Windt H, Mueller M, Badorrek P, Haefner D, Framke T, Koch A, Ziehr H, Krug N, Koch W, Hohlfeld JM. Safety, efficacy and repeatability of a novel house dust mite allergen challenge technique in the Fraunhofer allergen challenge chamber. Allergy. 2016 Dec;71(12):1693-1700. doi: 10.1111/all.12947. Epub 2016 Jun 23. PMID 27255590